CLINICAL TRIAL: NCT03246425
Title: Influence of Mechanical Ventilation Mode on Arterial Pressure Variations- a Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 909804-2
Record Dates: First submitted 2017-02-02; First posted 2017-08-11 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2017-08

CONDITIONS: Blood Pressure; Critical Illness; Hypovolemia
MeSH Terms: conditions — Critical Illness; Hypovolemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- 1. Volume control- Pressure control- APRV- VPA group (Active Comparator)
  Interventions: Other: Ventilator mode change; Device: Monitoring of blood pressure variation
- 2. Pressure control- APRV- Volume control- PAV group (Active Comparator)
  Interventions: Other: Ventilator mode change; Device: Monitoring of blood pressure variation
- 3. APRV- Volume control- pressure control- AVP group (Active Comparator)
  Interventions: Other: Ventilator mode change; Device: Monitoring of blood pressure variation

INTERVENTIONS:
Other: Ventilator mode change — The enrolled subjects will be moved from the baseline mode to another mode of ventilation and the changes in the arterial pulse will be observed
Device: Monitoring of blood pressure variation — The changes in the blood pressure will be measured in the form of Stroke Volume Variation using SVV using Vigileo (Edward Life sciences) monitor

SUMMARY:
Mechanical ventilation has been known to produce changes in the flow of blood through the major blood vessels in the body. These changes may go undetected, but with continuous arterial blood pressure measurements, changes in the arterial waveform can be visualized. Although we know that these arterial pressure variations occur during mechanical ventilation, little is known about the effects of various modes of mechanical ventilation on these changes. The most common modes of ventilation used in ICU are Volume control, Pressure control and Airway pressure release ventilation.

Objective We have designed a prospective randomized pilot study to determine the effects of the commonly used ventilator modes on the arterial pressure.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 yrs of age and older, Patients on mechanical ventilation, Patients deeply sedated in the ICU with RASS scores of atleast -3, Patients having an A-line for blood pressure monitoring, Patients with stable hemodynamics.

Exclusion Criteria:

Patients with moderate-severe ARDS, Patients requiring high inspiratory oxygen requirements, High peak inspiratory pressures requirement for ventilation, Presence of arrhythmia, Patients with spontaneous breathing activity, Patients on weaning mode, Patients having CHF or Cor pulmonale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
The study is to compare the effects of different modes of mechanical ventilation on arterial pressure variations. The arterial pressure variations will be measured as changes in the Stroke Volume Variation. | For 12 months
The study is to compare the effects of different modes of mechanical ventilation on arterial pressure variations. The arterial pressure variations will be measured as changes in the Pulse Pressure Variation | 12 Months

SECONDARY OUTCOMES:
Secondary outcome measured will be the influence of Airway Pressure Release Ventialtion (APRV) on arterial pressure measured using Pulse Pressure Variation | For 12 months
Secondary outcome measured will be the influence of Airway Pressure Release Ventialtion (APRV) on arterial pressure measured using Stroke Volume variation. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlos J Lopez, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States